CLINICAL TRIAL: NCT06674889
Title: Cancer Survival and Outcomes Impact of Universal Disability Screening and Cancer Rehabilitation Referral Among Adults With Cancer Referred to the University of North Carolina
Brief Title: Rehabilitation Outcomes Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2340
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Malignant Tumor
Keywords: rehabilitation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (No Intervention): Subjects will receive standard of care.
- Rehabilitation (Experimental): Subjects will be assessed for rehabilitation and a rehabilitation plan will be generated.
  Interventions: Other: Rehabilitation-based intervention

INTERVENTIONS:
Other: Rehabilitation-based intervention — Assessment of the subject by a specialty consultation and exercise program development.
  Arms: Rehabilitation

SUMMARY:
This pilot health services interventional study aims to prospectively assess the effectiveness of a pre-treatment rehabilitation (prehabilitation) program across a diverse cohort of adult cancer patients via a randomized pilot trial. Upon screening and identification of high-risk features through a central navigation process, patients referred to oncology clinics will be approached to participate in tailored prehabilitation interventions. The study will track and analyze functional outcomes and quality of life aiming to demonstrate the comprehensive benefits of prehabilitation on the cancer treatment continuum. We hypothesize that this referral program is feasible and that those randomized to the intervention arm will have superior functional outcomes and global health-related quality of life.

The rationale for this study is anchored in the urgent need to optimize the cancer care trajectory for high-risk patients whose treatment outcomes and quality of life are jeopardized by the multifaceted challenges of their disease. While prehabilitation has shown potential to mitigate these adverse effects, the optimal methods for identifying and connecting these high-risk individuals to appropriate prehabilitation resources remain underexplored. This study, with its systematic approach to enrolling a diverse adult cancer population, endeavors to investigate not only the benefits of prehabilitation interventions but also the effectiveness of a targeted referral process. By doing so, it aims to uncover novel strategies for efficiently allocating prehabilitation resources, thereby enhancing the precision and impact of supportive cancer care.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained to participate in the study and HIPAA authorization for the release of personal health information.
* Subjects are willing and able to comply with study procedures based on the judgement of the investigator.
* Age ≥ 18 years at the time of consent.
* The subject has been screened by the Central Oncology Navigation Program and referred to cancer care at the University of North Carolina Medical Center.
* Answer "yes" to at least one of the following screening questions:

  1. Does your health interfere with any of your activities of daily living (ADLs)?
  2. Have you fallen, or do you feel unsteady while standing or walking?
  3. Do you use durable medical equipment (DME)?
  4. Are you interested in increasing the amount you exercise?

Exclusion Criteria:

* Inability to read and understand the English language.
* Psychological or other disability resulting in the inability to provide informed consent.
* Unstable medical comorbidity that precludes safe participation in an exercise program, in the judgment of the clinical investigator.
* Prisoners and other institutionalized individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The proportion of rehabilitation interventions accepted | Baseline
  The proportion of pre-treatment rehabilitation intervention performed for patients who are referred to cancer rehabilitation and attend an initial appointment.

SECONDARY OUTCOMES:
Satisfaction rate | Baseline and post-3 months
  Acceptability in the subjects randomized to the intervention arm will be defined by the proportion of participants who report being "Neutral," & amp;#34; "Satisfied& amp;#34;" or & amp;#34;"Very Satisfied"& amp;#34; with the intervention utilizing the Experience with the Rehabilitation Program questionnaire.
  The questionnaire has 8 questions measured on a 5-point Likert scale: Not Effective At All=0, Slightly Effective=1, Moderately Effective=2, Very Effective =3, Extremely Effective =4. Minimum score= 0, maximum score=32.
Differences in physical function | Baseline and post-3 months
  Differences in physical function in the cancer rehabilitation arm and standard of care arm will be determined using PROMIS Short Form v2.0 Physical Function 4a. The PROMIS Short Form v2.0 - Physical Function 4a is a self-reported measure designed to assess an individual's capability to perform physical activities rather than their actual performance. The form consists of 4 items, each rated on a 5-point Likert scale ranging from "Without any difficulty" to "Unable to do." The scores are then summed to provide a total score, which can be converted to a T-score for standardized interpretation. The T-score has a mean (average) of 50 and a standard deviation of 10. A higher T-score indicates better physical function. Conversely, a lower T-score indicates poorer physical function.
Differences in participant activation | Baseline and post-3 months
  Differences in participant activation in the cancer rehabilitation arm and standard of care arm will be determined using Patient Activation Measure (PAM) 10 (Patient Activation Measure 10) scores. The Patient Activation Measure (PAM) 10 is a validated questionnaire designed to assess an individual's knowledge, skills, and confidence in managing their own health and healthcare. It consists of 10 items that measure patient activation, which is the extent to which individuals feel capable of managing their health. The PAM 10 includes 10 statements that respondents rate based on their level of agreement, ranging from "Strongly Disagree" to "Strongly Agree." Responses are scored on a scale from 0 to 100. Higher scores indicate greater patient activation.
Differences in overall health | Baseline and post-3 months
  Differences in overall health in the cancer rehabilitation arm and standard of care arm will be determined using PROMIS Global Health (PROMIS Scale v1.2 Global Health) scores. The PROMIS Global Health (PROMIS Scale v1.2 Global Health) is a comprehensive tool designed to assess an individual's overall physical, mental, and social health. The PROMIS Global Health v1.2 includes 10 items that cover various health domains. These items are divided into two main components: Global Physical Health and Global Mental Health. Global Physical Health: This includes items related to physical functioning, pain, fatigue, and overall physical health. Global Mental Health: This includes items related to mental health, emotional distress, and social health.Response Options: Each item is rated on a 5-point Likert scale, with higher scores indicating better health.Raw Scores: The responses are summed to create raw scores for both the Global Physical Health and Global Mental Health components. T-Scores: Th
Differences in physical activity levels | Baseline and post-3 months
  Differences in physical activity levels in the cancer rehabilitation arm and standard of care arm will be determined using the Godin Physical Activity Questionnaire (Godin-Shephard Leisure-Time Physical Activity Questionnaire)(GSLTPAQ)) scores. GSLTPAQ is used to assess an individual's physical activity levels during their leisure time. It focuses on the frequency and intensity of physical activities performed over a typical 7-day period.
  The questionnaire asks the number of times per week they engage in three types of physical activities for more than 15 minutes: Strenuous, Moderate, and Light Exercises. Strenuous exercise examples are running, vigorous swimming, and soccer), moderate exercise examples are fast walking, easy swimming, and volleyball, light exercise examples are yoga, easy walking, and bowling. Scoring: The responses are used to calculate a Leisure Score Index (LSI), which quantifies the total w
Overall survival | Up to one year
  Overall survival is defined from enrollment to death from any cause and obtained via medical record abstraction.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E Jensen, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- The N.C. Cancer Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Data could be available on request, though there is no plan to store data in any kind of publicly available repository.